CLINICAL TRIAL: NCT00219869
Title: Galantamine in the Preventive Treatment of Chronic Post-Traumatic Headache
Brief Title: Galantamine in the Treatment of Post-Traumatic Headache
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rapoport, Alan, M.D. (Individual)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAL-EMR-4006
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Post-Traumatic Headache; Head Trauma,Closed; Retention Disorders,Cognitive
Keywords: Post; Traumatic; Headache; Cognitive
MeSH Terms: conditions — Post-Traumatic Headache; Head Injuries, Closed; Memory Disorders; Headache | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine

SUMMARY:
Most patients with CPTH present with additional major cognitive, behavioral and somatic problems. Most drugs used currently have a negative influence on cognition. Therefore, treatment strategies addressing both the headache and cognitive disturbances in patients with CPTH are necessary. (CPTH; Chronic Post Traumatic Headache).

DETAILED DESCRIPTION:
Headache is the most common symptom after a closed head injury, persisting for more then 2 months in 60% of the patients. CPTH is an important cause of consultations in neurology offices and headache clinics, posing a severe burden and affecting the quality of life of sufferers.

ELIGIBILITY:
Inclusion Criteria:

Age range 18-75 CPTH according to ICHD-2 Fertile woman using adequate birth control Willing and able to give informed consent Willing and able to complete the entire course of the study to comply with study instructions Stable does of preventive medication

-

Exclusion Criteria:

Subject is pregnant or lactating Significant medical or psychiatric disease Previous failure to 4 or more adequate trials of preventive medication Patient on non-stable dose of medication used to prevent CPTH

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-07; Study Completion 2005-08

PRIMARY OUTCOMES:
Primary Headache Efficacy Measure; number of pain free days after 3 months

SECONDARY OUTCOMES:
Consumption of rescue medication
Number of days with moderate or severe headache after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Rapoport, MD, Principal Investigator — The New England Center for Headache
Locations (1):
- The New England Center for Headache, Stamford, Connecticut, United States